CLINICAL TRIAL: NCT01415609
Title: Establishment of Registry for Endoscopic Submucosal Dissection for Superficial Gastrointestinal Neoplasia
Brief Title: Endoscopic Submucosal Dissection Registry
Acronym: ESD Registry
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Olympus (Industry)
Responsible Party: Michael B Wallace, MD, MPH, Mayo Clinic Florida
Other Study IDs: 10-000160
Record Dates: First submitted 2011-08-10; First posted 2011-08-12 (Estimated); Last update posted 2012-11-09 (Estimated); Status verified 2012-11

CONDITIONS: Gastrointestinal Neoplasms; Gastric Cancer
Keywords: Gastrointestinal neoplasia; Submucosal resection
MeSH Terms: conditions — Gastrointestinal Neoplasms; Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to monitor the success rates and completion rates for endoscopic submucosal dissection (ESD) for gastrointestinal (GI) cancers.

ELIGIBILITY:
Inclusion Criteria: Patients referred for endoscopic treatment of advanced gastrointestinal (colorectal, gastric, duodenal, esophagus) neoplasia, defined by any of the following procedures:

1. Flat dysplastic lesion greater than 2cm(IIa or IIb by Paris classification)
2. Flat depressed lesion < 2cm in size (llc by Paris Classification)
3. Ulcerated lesion < 2cm (Paris type lll) staged as T1N0 on endoscopic ultrasound
4. Upon resection, the criteria for curative ESD include:

   * Non-invasive neoplasia of differentiated carcinoma
   * No lymphovascular invasion
   * Intramucosal cancer or minute submucosal cancer <1 mm invasion (sm1)
   * Negative deep and lateral margins.

Exclusion Criteria:

1. Use of antiplatelet(e.g. clopidrogel) or anticoagulation (e.g. Coumadin) agents that cannot be withheld for at least 7 days prior to the procedure. Aspirin use is accepted according to the American Society for Gastrointestinal Endoscopy for these procedures.
2. Patients who refuse or who are unable to consent.
3. Suboptimal colon prep, or solid gastric residual that precludes safe lesion resection at the time of endoscopy.
4. Lesion location in a segment of the colon not conducive to ESD, including significant narrowing, tortuosity and/or extensive diverticular disease, as determined by the endoscopist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred for endoscopic treatment of gastrointestinal neoplasia.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2010-08; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Ease of use of the overall procedure and Time of procedure. | 1 Year
  * Ease of use of overall procedure as rated on a 5-point visual analog scale for very easy, easy, neutral, difficult and very difficult.
  * Time (in minutes) needed to resect the lesion completely, as measured from the first injection to final excision of the lesion.

SECONDARY OUTCOMES:
Complications and Rate of Completion | 1 Year
  * Minor and Major Bleeding
  * Minor and Major perforation
  * Post-polypectomy syndrome (defined as the presence of moderate or severe pain persisting more than 2 hours following completion of the procedure).
  * Other(any other adverse event which the investigator feels is potentially attributable to the procedure).
  * Enbloc resection of all endoscopically visible neoplasia
  * Pathologically negative for lateral and/or deep margins
  * Absence of residual neoplasia confirmed by repeat standard colonscopy and biopsy of ESD site 3-6 months following the index procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Wallace, MD,MPH, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Florida, Jacksonville, Florida, United States